CLINICAL TRIAL: NCT04622826
Title: Studio in Aperto Sulla Somministrazione di Plasma di Paziente Convalescente da COVID- 19 a Paziente Con Polmonite COVID-19 Ospedalizzato, Non in Terapia Intensiva
Brief Title: plasmApuane CoV-2 : Efficacy and Safety of Immune Covid-19 Plasma in Covid-19 Pneumonia in Non ITU Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Responsible Party: Principal Investigator, mirko lombardi, consultant, Azienda USL Toscana Nord Ovest
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ATNONordOvest
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Covid-19 Pneumonia
Keywords: covid-19 pneumonia; convalescent plasma; hyperimmune plasma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sequential immune plasma infused patients (Experimental): immune covid 19 plasma infusion
  Interventions: Biological: immune plasma

INTERVENTIONS:
Biological: immune plasma — immune covid 19 plasma infusion

SUMMARY:
Aim of the study is to verify the efficacy and safety of convalescent hyperimmune plasma infusion in hospitalized covid-19 patients non in ITU with pneumonia and respiratory symptoms within seven days from the beginning of symptoms.

Efficacy is evaluated by the number of patients who will improve their clinical condition and will not be admitted to ITU. .Safety is considered in relation to adverse reactions to plasma infusion.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* hospitalized patients with positive covid-19 swab with respiratory symptoms and CT confirmation of covid-19 chest disease admitted to non ITU recovery area.
* informed consent for plasma infusion
* informed consent to blood samples storing for future studies.

Exclusion Criteria:

* pregnant or breastfeeding female patient or planning for a pregnancy in the period of the study

  * immunoglobulin infusion in the last month

contraindication to transfusion or previous adverse reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
ITU admission | up to 30 days
  number of patients admitted to ITU after immune plasma transfusion
administration of O2 | up to 30 days
  O2 support will be monitored and reported in its various modes of administration (e.g. nasal cannula, high flow nasal cannula, noninvasive ventilation, mechanical ventilation)
hospital mortality | up to 90 days
  number of subject deaths
immune plasma infusion adverse reaction | in the first 24-48 hours
  number of participants with treatment-related adverse events as assessed by CTCAE v4.0"

CONTACTS AND LOCATIONS:
Overall Officials: antonella vincenti, Principal Investigator — ospedale delle Apuane
Locations (1):
- Ospedale delle Apuane, Massa, Tuscany, Italy